CLINICAL TRIAL: NCT03436914
Title: Treatment Response of Maintenance Dose of Proton Pump Inhibitor in Patients With Nonerosive Gatroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-1143
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Non-erosive Gatroesophageal Reflux Disease

STUDY DESIGN:
Intervention Model Description: There is only one arm in this study. Patients diagnosed as NERD will take PPI (Esomezol) for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PPI (Experimental): Esomezol®
  Interventions: Drug: PPI

INTERVENTIONS:
Drug: PPI — After the diagnosis of NERD through patient's symptom and endoscopy, PPI (esomezol) will be given for 8 weeks. The effect of PPI for NERD patients will be analyzed.
  Other Names: Esomezol®

SUMMARY:
For ERD(erosive reflux disease), which pathogenesis is mainly the acid reflux mechanism, primary treatment is therefore PPI. However, NERD(non-erosive reflux disease) is much more complex than ERD and there are more factors causing the typical symptoms. As a result, there is no consensus for the treatment of NERD besides using PPI similar to GERD(gastroesophageal reflux diseas). This study intent to evaluate the effect of PPI(Esomezol) on NERD patients and analyze the improvement of symptoms and the factors related to the result.

DETAILED DESCRIPTION:
(1) Among GERD patients, EGD(esophagogastroduodenoscopy) must be done before 6 months and must prove there is no erosive lesion. (2) During EGD, esophagus mucosa histology will be taken for evaluation. (3) For NERD patients, Esomezol is given once a day (before breakfast meal), for whole 8 weeks. (4) PAGI-SYM and HAD-K is evaluated and score just before the administration of PPI, 4weeks after and 8weeks after the study initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 19 years old
* Patient with typical GERD symptom (heartburn or acid reflux more than once a week)

Exclusion Criteria:

* Patient who received EGD since the past 6 months, and diagnosed as GERD endoscopically
* Patient with active gastric/duodenal ulcer
* Patient who received esophagus, stomach or duodenum surgery
* Patient with hypersensitivity to esomezol®
* Patient with no achieved agreement on the study from the guardian or patient himself.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Proportion of PAGI-SYM score (0-2) patients after 8 weeks of PPI(Esomezol) | 8 weeks
  Scoring the PAGI-SYM to analyze the satisfaction of symptoms (heartburn and regurgitation) after 8 weeks of PPI administration to NERD patients

SECONDARY OUTCOMES:
The analysis of factors affecting the PAGI-SYM inculding immunolgic array and esophagus mucosal microbiota | 8 weeks
  The analysis of complete symptom (regurgitation, heartburn) remission (PAGI-SYM score 0) after 8weeks of PPI

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No